CLINICAL TRIAL: NCT06914050
Title: An Exploratory Study on the Treatment of Limited-stage Small Cell Lung Cancer With Induction Therapy of Adebrelimab Combined With Chemotherapy Followed by Thoracic Radiotherapy After Hypofractionated Radiotherapy
Brief Title: Hypofractionated Radiotherapy Followed by Chemo-immunotherapy Induction Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS-SCLC
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer, Small Cell; Limited-stage Small Cell Lung Cancer (LS-SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): SERT+Chemo-immunotherapy+CCRT+Immunotherapy maintenance
  Interventions: Drug: Adebrelimab; Drug: EC/EP; Radiation: SBRT; Radiation: Chest radiotherapy

INTERVENTIONS:
Drug: Adebrelimab — Induction therapy：Adebrelimab, 1200mg, d1, q3w, 2 cycles; Maintenance therapy：Adebrelimab, 1200mg, d1, q3w, until disease progression or unbearable toxicity.
Drug: EC/EP — Chemotherapy: standard chemotherapy EC/EP
Radiation: SBRT — 8Gy*3
Radiation: Chest radiotherapy — Chest radiotherapy: conventional fractionation mode 2Gy QD total dose 60Gy or 1.5Gy BID total dose 45Gy, according to the patient's physical condition, concurrent EP or EC chemotherapy can be considered

SUMMARY:
Radiotherapy can activate local and systemic immune responses through a variety of mechanisms, which can enhance anti-tumor immune effects. The dose fractionation pattern of radiotherapy has an important influence on the occurrence of immune-induced effects. Stereotactic body radiation therapy (SBRT) has obvious advantages in activating interferon effects and inducing abscopal effects. SBRT combined with immunity can enhance the abscopal effect induced by radiotherapy and play a synergistic role. The 8Gy×3 fractionation scheme is currently the most widely used stereotactic radiotherapy scheme. Because we conducted this study, the primary lesion received large-fraction partial tumor irradiation and then received adebrelimab combined with chemotherapy induction treatment for 2 cycles, followed by sequential chest radiotherapy for the treatment of limited-stage small cell lung cancer, to explore the effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old; 2. Limited-stage small cell lung cancer (AJCC 8th) confirmed by histology or cytology; 3. Subjects have not received any treatment for SCLC; 4. Have measurable target lesions according to RECIST v1.1; 5. ECOG score of 0-1; 6. Life expectancy ≥ 12 weeks; 7. Normal function of major organs, that is, meet the following criteria:

1. Routine blood tests must meet the following criteria (no blood transfusion, no use of hematopoietic factors, and no use of drug correction within 14 days):

   1. ANC ≥ 1.5×109/L;
   2. PLT ≥ 100×109/L;
   3. HB ≥ 90 g/L;
2. Biochemical tests must meet the following criteria:

   1. TBIL ≤ 1.5×ULN;
   2. ALT, AST≤ 2.5×ULN;
   3. Serum creatinine sCr≤1.5×ULN, endogenous creatinine clearance ≥50mL/min (Cockcroft-Gault formula);
3. Coagulation function must meet the following requirements: INR≤1.5×ULN and APTT≤1.5×ULN; 8. Female subjects of childbearing age must undergo a serum pregnancy test within 3 days before starting the study medication, and the result must be negative, and they must be willing to use a medically approved high-efficiency contraceptive measure (such as intrauterine contraceptive device, contraceptive pills or condoms) during the study and within 3 months after the last administration of the study medication; for male subjects whose partners are female subjects of childbearing age, they must be surgically sterilized or agree to use an effective contraceptive method during the study and within 3 months after the last administration of the study medication.

9. The subjects voluntarily join this study, sign the informed consent form, have good compliance, and cooperate with follow-up visits.

Exclusion Criteria:

1. Central nervous system metastasis;
2. Any active autoimmune disease or history of autoimmune disease (including, but not limited to: moderate interstitial pneumonia and above, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis; patients with vitiligo or childhood asthma that has completely resolved and does not require any intervention as an adult can be included; patients who require bronchodilators for medical intervention are not included;
3. Patients with congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/mL), hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the detection limit of the analytical method) or co-infection with hepatitis B and hepatitis C, active pulmonary tuberculosis;
4. Immunosuppressive drugs have been used within 14 days before the first use of study drugs, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroid hormones (i.e. no more than 10 mg/day prednisone or its equivalent);
5. Vaccination with live attenuated vaccine within 4 weeks before the first dose or planned during the study;
6. Suffering from other malignant tumors in the past 3 years;
7. Evidence of past or current pulmonary fibrosis, interstitial pneumonia (grade II or above), pneumoconiosis, radiological pneumonia, drug-induced pneumonia, and severe lung function impairment;
8. Uncontrolled hypertension;
9. Suffering from myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including QTc interval ≥450ms for males and ≥470ms for females). According to NYHA standards, patients with grade III-IV heart failure, or left ventricular ejection fraction (LVEF) <50% indicated by cardiac ultrasound examination, had myocardial infarction within 6 months before enrollment, New York Heart Association grade II or above heart failure, uncontrolled angina pectoris, uncontrolled severe ventricular arrhythmias, clinically significant pericardial disease, or ECG indicating acute ischemia or abnormal active conduction system;
10. Severe infection within 4 weeks before the first medication (such as: intravenous infusion of antibiotics, antifungal or antiviral drugs for more than 7 days), or unexplained fever >38.5°C during the screening period/before the first medication;

1 1. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 12. Pregnant or lactating women; patients with fertility who are unwilling or unable to take effective contraceptive measures; 13. Known to have allergic reactions, hypersensitivity reactions or intolerance to adebrelimab (SHR-1316), etoposide, cisplatin or its excipients; 14. Subjects who are participating in other clinical studies or whose first medication time is less than 4 weeks from the end of the previous clinical study (last medication) or 5 half-lives of the study drug; 15. Subjects with a history of psychotropic drug abuse, alcoholism or drug abuse; 16. The researcher believes that there are any conditions that may harm the subject or cause the subject to be unable to meet or perform the study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival | 24months

SECONDARY OUTCOMES:
Objective response rate | 24months
Overall survival | 24months
TRAEs | 24months

IPD SHARING:
Plan to Share IPD: No